CLINICAL TRIAL: NCT02896673
Title: Evaluation of the Diagnostic Performance of Electrical Impedance Tomography (EIT) to Detect Situations at Risk of Lesions Induced by Conventional Mechanical Ventilation in Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Evaluation of the Diagnostic Performance of Electrical Impedance Tomography to Detect Situations at Risk of Lesions Induced by Conventional Mechanical Ventilation in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-642
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Distress Syndrome
Keywords: positive expiratory pressure (PEP); Acute Respiratory Distress Syndrome (ARDS); electrical impedance tomography (EIT); tidal volume (TV); transpulmonary pressure (TPP)
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Weights and Measures

ARMS (1):
- ventilatory conditions and measures with scanner and EIT (Experimental): The patient is installed on the scanner bed, EIT electrodes are connected to the acquisition device of the EIT signal.
  Esophageal pressure signals, pressure and flow in the airways will be acquired continuously
  Interventions: Procedure: ventilatory conditions and measures with scanner and EIT

INTERVENTIONS:
Procedure: ventilatory conditions and measures with scanner and EIT — Different ventilatory conditions are studied and measures are acquired with scanner and EIT
  Time A: measure under basal conditions (TVbasal=6ml/kg of predicted weight), basal PEP, basal inspiratory time / total time = 30%)
  Time B: different PEP are applied for 4 minutes: 5, 10, 15, 20 cm of H2O conserving the basal TV
  Time C: different TV are applied for 4 minutes: 4, 7, 10 ml/kg of predicted weight conserving the basal PEP and the basal inspiratory time
  Time D: recruitment in continuous positive airway pressure at 45 cm of H2O is performed for 30 seconds
  Time E: return to adjustment period A

SUMMARY:
Acute respiratory distress syndrome remains a serious condition, with a mortality rate of between 30 and 50%. The use of mechanical ventilation with small tidal volumes, and by limiting the plateau pressure in the respiratory tract below 30 cm H2O has been shown to reduce mortality by approximately 10%, probably by reducing pulmonary hyperinflation and pulmonary lesions induced by mechanical ventilation. It is therefore now established that the respirator settings influence patient prognosis. However, around 30% of patients with ARDS ventilated with these settings supposedly protective continue to present signs of pulmonary hyperinflation on tomodensitometry, suggesting an additional reduction in the tidal volume could be required in certain patients. Electrical impedance tomography (EIT) is a new imaging technique that gathers functional pulmonary information at bedside.

This technique also allows a regional analysis, allowing the complexity of the spatial distribution of ARDS pulmonary lesions to be understood. The hypothesis is that EIT is a reliable method to detect at-risk situations of lesions induced by mechanical ventilation among patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Hospitalised in the medical resuscitation department of the Croix Rousse hospital, Lyon, Fr
* With ARDS according to the 1994 American-European Consensus Conference
* Duration of ARDS less than 96 hours
* With invasive mechanical ventilation
* With sedative and analgesic treatment for adaptation of the respirator with or without neuromuscular blocking agents
* Consent obtained from patient family
* Indication for thoracic scanner as judged by the physician in charge of the patient

Exclusion Criteria:

* Excessively serious respiration precluding the modifications to ventilation planned in the protocol

  * severe hypoxemia defined as sever by arterial blood pressure/fraction of inspired oxygen (PaO2/ FiO2) below 100 mm Hg in dorsal decubitus position
  * uncontrolled respiratory acidosis, defined by a pH below 7.25, despite an increase of respiratory frequency up to 35/min and a tidal volume up to 8 mL/kg of predicted weight
  * respiratory system plateau pressure higher than 30 cm H2O, with a tidal volume below or equal to 6 mL/kg of predicted weight.
* Contraindication for transport to the radiology department

  * uncontrolled hemodynamic instability defined by a mean arterial blood pressure below 65 mm Hg, despite use of antihypotensive agents
  * patient requiring continuous dialysis without possibility for disconnection for reason of uncontrolled metabolic acidosis (pH<7.20).
* Without reliable monitoring during transport of the patient to the radiology department

  * absence of invasive arterial pressure measurement
  * unreliable measurement of arterial saturation in oxygen (SpO2) defined by a perfusion index below 0.5.
* Intracranial hypertension
* Impossible to apply EIT electrodes on the thorax of the patient (burns, dressings, …)
* Undrained pneumothorax or bronchopleural fistula
* Scanner unavailable for the study (broken down, overloaded program, …)
* Contraindication esophageal balloon catheter

  * Known or suspected esophageal disease (tumor, esophageal varices, esophagitis, diverticulum, ...)
  * Latex allergy
* Patient previously included in the study
* Vulnerable persons (as defined in laws L1121-5 to L1121-7, L1121-8 and L1122-1-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2015-01-21 (Actual); Study Completion 2015-01-21 (Actual)

PRIMARY OUTCOMES:
mean values of optimal PEP obtained by EIT | after 2 minutes of applying each ventilatory experience
  Data acquisition will be carried out for 2 minutes and will start after 2 minutes of applying each ventilatory long time experience (A, B, C, E).
  mean values of optimal PEP will be compared between the 2 methods (scan and EIT).
mean values of optimal TV obtained by EIT | after 2 minutes of applying each ventilatory experience
  Data acquisition will be carried out for 2 minutes and will start after 2 minutes of applying each ventilatory long time experience (A, B, C, E).
  mean values of optimal TV will be compared between the 2 methods (scan and EIT)
mean values of optimal PEP obtained by scan | after 4 minutes of applying each ventilatory experience
  Data acquisition will start after 4 minutes of applying each ventilatory long time experience (A, B, C, D).
  mean values of optimal PEP will be compared between the 2 methods (scan and EIT).
mean values of optimal TV obtained by scan | after 4 minutes of applying each ventilatory experience
  Data acquisition will start after 4 minutes of applying each ventilatory long time experience (A, B, C, D).
  mean values of optimal TV will be compared between the 2 methods (scan and EIT).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France